CLINICAL TRIAL: NCT03132519
Title: Optimal Remifentanil Site-effect Concentration for Preventing Severe Cough and Hyperdynamic Response During Tracheal Extubation After Sevoflurane vs. Desflurane. A Randomized Clinical Trial
Brief Title: Optimal Remifentanil Ce for Preventing Severe Cough and Hyperdynamic Response During Tracheal Extubation
Acronym: REX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Principal Investigator, Fredy Ariza, Anesthesiologist, Fundacion Clinica Valle del Lili
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REX
Record Dates: First submitted 2014-04-25; First posted 2017-04-28 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Cough; Hypertension
Keywords: Cough; Hypertension; Remifentanil; Sevoflurane; Desflurane
MeSH Terms: conditions — Cough; Hypertension | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Sevo-2.0 (Experimental): This group will maintain remifentanil infusion by TCI to 2 ng/ml during emergence and extubation after have received sevoflurane during procedure.
  Interventions: Drug: Remifentanil
- Sevo-2.5 (Experimental): This group will maintain the remifentanil infusion by TCI to 2.5 ng/ml during emergence and tracheal extubation after have received sevoflurane during surgical procedure.
  Interventions: Drug: Remifentanil
- Des-2.0 (Experimental): This group will maintain the remifentanil infusion by TCI to 2.0 ng/ml during emergence and tracheal extubation after have received desflurane during surgical procedure.
  Interventions: Drug: Remifentanil
- Des-2.5 (Experimental): This group will maintain the remifentanil infusion by TCI to 2.5 ng/ml during emergence and tracheal extubation after have received desflurane during surgical procedure.
  Interventions: Drug: Remifentanil
- Sevo-Control (Active Comparator): This group will maintain the remifentanil infusion by TCI to 1.0 ng/ml during emergence and tracheal extubation after have received sevoflurane during surgical procedure.
  Interventions: Drug: Remifentanil
- Des-Control (Active Comparator): This group will maintain the remifentanil infusion by TCI to 1.0 ng/ml during emergence and tracheal extubation after have received desflurane during surgical procedure.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — To maintain remifentanil Ce at 1.0 (control) vs. 2.0 vs. 2.5 ng/ml by a TCI system during anesthesia emergence until tracheal extubation
  Other Names: Ultiva

SUMMARY:
Pain, cough, hypertension and tachycardia are frequent events during extubation due to a secondary stimulation of mechanoreceptors located in the airway. The mechanical effect of the endotracheal tube activates autonomic reflexes, a situation that could potentially impair the clinical condition of patients. Previous studies have used remifentanil during emergence and extubation showing good results to control this reflex response. However, it is unknown so far, the optimal effect site concentration (Ce) of remifentanil to allow a better control of these events with a low incidence of adverse effects after have received inhaled anesthesia plus remifentanil for anesthetic maintenance. This study will determine the Ce of remifentanil associated with a lower proportion of cough and hyperdynamic circulatory response during extubation for emergency after exposure to sevoflurane or desflurane.

DETAILED DESCRIPTION:
Single-center, randomized, double-blind protocol. The investigators aim to include 368 patients under balanced anesthesia with sevoflurane or desflurane to be randomly allocated into 6 different remifentanil Ce groups [77 individuals in each of interventional groups (2.0 vs. 2.5 ng/ml) and 30 in each of the control groups (1.0 ng/ml) administrated by a target-controlled infusion (TCI) system during emergence and tracheal extubation .

Once informed consent is obtained and inclusion/exclusion criteria are met, subjects will be randomized before starting of the surgical procedure. This information will remain blinded to the attendant anesthesiologist and the independent evaluator during the process of extubation, except for type of inhaled anesthetic for maintenance .

The intervention will start when the anesthesiologist decide to suspend the sevorane or desflurane dial. At this moment, the fresh flow gas of the anesthesia machine will be adjusted to 7-8 liters per minute and the infusion of remifentanil will be set up to establish a Ce of 2.0 ng/ml or 2.5 ng/ml. All patients will be extubated only when all of these three parameters exist: response to name by eyes opening, response to orders of breathing and mouth opening.

The evaluation and outcomes measurement will include: Presence and intensity of cough and changes in heart rate and blood pressure during eyes opening in response to calling by name, tracheal extubation and 2.5 min after, time to get to be extubated after inhaled anesthetic discontinuation, episodes of hypoxemia and sedation state during the first 25 minutes after extubation, requirements of rescue analgesia and postoperative nausea and vomit during this period.

Close monitoring of patients will take place and data will be collected during the preoperative, intraoperative and postoperative stages until discharge from the post anesthesia care unit. Lost to follow and adverse events will be assessed. An interim committee will evaluate partial results of the study when it reaches 25 and 50% of recruitment, so the investigators can continue building thereof according to analysis obtained.

Statistical analysis will be performed by a independent statistician based on "intention to treat" principle. In addition, excluded data and its reasons for exclusion will be evaluated. For the descriptive exploratory analysis, continuous variables will be presented as means (standard deviation) or medians (interquartile ranges). The degree of dispersion, shape and position as the fulfillment of normality will be analyzed using the t of Student or Mann-Whitney tests as appropriate. Categorical variables will be presented as proportions and compared using the chi-square or Fisher 's exact tests as appropriate. Time-varying measures analysis of variance for repeated measures will be used to make comparisons between groups.

ELIGIBILITY:
Study Population:

Patients undergoing planned surgery who want to avoid coughing during emergence and extubation (Head and Neck Surgery, abdominal, neurosurgery and intraocular)

Inclusion Criteria:

* American Society of Anesthesia status I and II
* Age between 18 to 60 years.
* Elective surgery.

Exclusion Criteria:

* Uncontrolled hypertension. (SBP> 180 mmHg) at pre anesthesia area.
* Active or uncontrolled pulmonary disease.
* Signs or history of difficult airway.
* Recent respiratory infection.
* Train-of-four (TOF) index <90% at the end of surgery.
* Patients who have received some form of pre oral medication.
* Body mass Index above 30 kg/m2.
* Concomitant use of epidural catheter.
* Urgent surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 364 (Actual)
Dates: Start 2013-10; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Cough during emergency from anesthesia | From eye opening up to 2.5 minutes after tracheal extubation
  Assess the presence and intensity of cough : 0) No cough, 1) A single episode of cough, 2) More than one episode of nonsustained cough, 3) sustained and repetitive cough with head elevation.

SECONDARY OUTCOMES:
Cardiac response during emergence from anesthesia | From discontinuation of inhalational anesthetics up to 2.5 minutes after tracheal extubation
  Assessment of heart rate (bpm) during awakening and tracheal extubation: Measurements of systolic blood pressure will be obtained at the time of suspending of the halogenated (Basal 2) , eye opening, tracheal extubation and 2.5 minutes after extubation
Pressor response during emergence from anesthesia | From discontinuation of inhalational anesthetics up to 2.5 minutes post-extubation
  Assessment of systolic blog pressure (mmHg) during awakening and tracheal extubation: Measurements of systolic blood pressure will be obtained at the time of suspending of the halogenated (Basal 2) , eye opening, tracheal extubation and 2.5 minutes after extubation
Time to eye opening | From inhaled anesthetic discontinuation until the moment of eye opening response to verbal command (calling by name), assessed up to 20 minutes.
  Time in seconds from inhaled anesthetic discontinuation to eye opening response to call by name and touch stimuli.
Time to tracheal extubation | From inhaled anesthetic discontinuation until the event of tracheal extubation, assessed up to 20 minutes.
  Time in seconds from inhaled anesthetic discontinuation to safety conditions for tracheal extubation (patients must respond positively to three different commands: "open your eyes " , "breath deep " and "open your mouth ")
Halogenated end tidal concentration at tracheal extubation | From eyes opening until the event of tracheal extubation, assessed up to 20 minutes.
  Inhaled gas concentration measured in vol % by the gas analyzer at tracheal extubation
Respiratory rate during post-extubation | From tracheal extubation to 25 minutes later
  Number of breaths per minute during spontaneous ventilation.
Post-extubation hypoxemia | From tracheal extubation to 25 minutes
  Continuous non-invasive measurement of the percentage of hemoglobin that is attached to oxygen through a pulse oximeter . Episodes of arterial oxygen saturation less than 92% , which is present in the next 10 minutes to extubation were recorded and encourage the patient to breathe through call and tactile stimulation as necessary during this time. If you arrived 10 minutes after extubation the patient continues to present desaturation because bradypnea / intermittent apnea the same process will continue until the patient has spontaneous ventilation ( breathing without any verbal or tactile stimulation ) .
Rescue analgesia requirement in the immediate postoperative time | From tracheal extubation up to first postoperative hour
  Amount of opioid requirements for rescue analgesia during first postoperative hour (other opioids dose will be converted to equipotent milligrams of morphine.
Postoperative nausea and vomiting | From tracheal extubation to first postoperative hour
  Rated on a scale of 0-3, representing presence and intensity of nausea and / or vomiting within the first postoperative hour 0 = no nausea
  1. = mild nausea without vomiting episodes
  2. = nausea and a single episode of vomiting
  3. = more than one episode of vomiting during the first hour

CONTACTS AND LOCATIONS:
Overall Officials: Fredy G Ariza, MD., MSc., Principal Investigator — Fundacion Clinica Valle del Lili; Ivan F Quintero, MD, Study Chair — Fundacion Clinica Valle del Lili
Locations (1):
- Fundacion Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Data available for future validations at institutional database system from Clinical Research Center, Fundación Valle del Lili of